CLINICAL TRIAL: NCT03058146
Title: A Novel Mobile Health Exercise Intervention in Aging: Brain Perfusion and Cognition
Brief Title: Independent Walking for Brain Health
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 shut down of research operations
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Zvinka Z. Zlatar, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20153238; K23AG049906 (NIH)
Record Dates: First submitted 2017-02-10; First posted 2017-02-20 (Actual); Results first posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Physical Activity; Aging
Keywords: Exercise; Fitness; Physical Activity; Cognitive Aging; Cerebral Blood Flow; Brain Imaging; Unsupervised Intervention; Mobile Health; Free-living exercise intervention
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial with ongoing enrollment into each arm (individual intervention)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Health Walking Condition (Experimental): Physically inactive older adults in this condition will perform 3 months of prescribed brisk walking (to increase cardio respiratory fitness) in their real world environments, using mobile health (mHealth) devices during each exercise session to achieve and maintain a minimum of 150 minutes of moderate to vigorous physical activity (MVPA) per week.
  Interventions: Behavioral: Mobile Health Walking Condition
- Healthy Aging Education Condition (Active Comparator): The education control condition will provide participants with printed materials and homework assignments on issues related to successful aging, such as nutrition, social activity, cognitive and social engagement.
  Interventions: Behavioral: Healthy Aging Education Condition

INTERVENTIONS:
Behavioral: Mobile Health Walking Condition — Physically inactive older adults in this condition will perform 3 months of prescribed brisk walking (to increase cardio respiratory fitness) in their real world environments, using mobile health (mHealth) devices during each exercise session to achieve and maintain a minimum of 150 minutes of moderate to vigorous physical activity (MVPA) per week.
  Arms: Mobile Health Walking Condition
Behavioral: Healthy Aging Education Condition — The education control condition will provide participants with printed materials and homework assignments on issues related to successful aging, such as nutrition, social activity, cognitive and social engagement.
  Arms: Healthy Aging Education Condition

SUMMARY:
Physical activity interventions with older adults can improve brain health; however most interventions have been performed in gym-like settings that reach a small sector of the senior population. Since not everyone can access a gym, it is important to study whether brisk walking in real world environments can also help brain health. This study will use mobile health devices to help older adults independently walk for brain health, thus representing a critical step towards the dissemination of physical activity intervention programs aimed at preserving cognitive function in aging.

DETAILED DESCRIPTION:
Physical activity interventions conducted in supervised settings (laboratories and group settings) with older adults have consistently shown improved cardiovascular and cerebrovascular health and improved cognitive function. What is lacking is the development of interventions that take place in real world environments and that take advantage of new technologies to help objectively track real time physical activity behaviors. Real world physical activity interventions have the potential to reach a larger segment of the population and to enhance maintenance after the intervention period ends. This study will develop a novel physical activity intervention using mobile health technologies to promote physical activity levels likely to affect cerebral blood flow and cognition in real world environments in cognitively normal older adults. A randomized controlled trial will be conducted with 30 participants being assigned to the mobile health physical activity condition (walking in free-living environments tracked via mobile health technologies) and another 30 to an education control condition (at home reading about healthy aging materials) for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 65-80
* Ability to obtain a signed physician's clearance for participation in this study
* English-speaking as needed to complete cognitive testing and follow study procedures
* Cognitively normal (based on comprehensive neuropsychological assessment)
* No contraindications for Magnetic Resonance Imaging (MRI)
* Must be ambulatory and able to walk independently

Exclusion Criteria:

* History of head injury involving loss of consciousness within the past 6 months and/or history of severe traumatic brain injury
* Major neurological disorders (dementia, multiple sclerosis, epilepsy, etc)
* Chronic major psychiatric disorders (schizophrenia, major recurrent affective disorder)
* History of major vascular events (myocardial infarction, stroke, etc),
* History of diabetes
* History of falls in the last year resulting in hospitalization
* Unstable or poorly controlled medical problems e.g. heart failure, diabetes (poorly controlled or on insulin), uncontrolled hypertension, pulmonary disease with hypoxia or hypercapnia, significant liver problems or renal failure, treatment of cancer in the past 2 years (other than non-melanoma skin cancer), HIV positive
* Objective evidence of cognitive impairment based on neuropsychological assessment

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zvinka Z Zlatar, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
Access to databases and associated software tools generated under the project will be available for educational, research and non-profit purposes. Such access will be provided using web-based applications, as appropriate. Publication of data shall occur during and at the end of the project, consistent with normal scientific practices. Research data which documents, supports and validates research findings will be made available after the main findings from the final research data set have been accepted for publication. Such research data will be redacted to prevent the disclosure of personal identifiers.

REFERENCES:
- [Derived] Hays Weeks CC, Moore AA, Allison M, Patrick K, Bondi MW, Nebeker C, Liu TT, Wing D, Higgins M, Hartman SJ, Rissman RA, Zlatar ZZ. The Independent Walking for Brain Health Intervention for Older Adults: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2023 Feb 13;12:e42980. doi: 10.2196/42980. PMID 36535765
- [Derived] Nebeker C, Zlatar ZZ. Learning From Older Adults to Promote Independent Physical Activity Using Mobile Health (mHealth). Front Public Health. 2021 Aug 12;9:703910. doi: 10.3389/fpubh.2021.703910. eCollection 2021. PMID 34476229

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ongoing studies at the University of California San Diego and the Shiley-Marcos Alzheimer's Disease Research Center, as well as from ResearchMatch, flyers, community engagement talks (ie, talks at retirement communities, senior centers, libraries, and health fairs) and by word of mouth. All participants were enrolled between October 2017 and March 2020, at which time study recruitment was terminated because of the COVID-19 pandemic.
Pre-assignment Details: 53 participants were enrolled (signed informed consent). After enrollment, 7 did not meet further eligibility criteria (based on cognitive and fitness testing) and 2 did not complete the baseline sessions due to the COVID-19 shut down. Out of 53 enrolled, 44 were randomized to the exercise (n=21) and control conditions (n=23). One participant randomized to the control condition could not start the intervention due to the COVID-19 shut down. Total analytic sample is N=43 (exercise=21,control=22).
Groups:
- Physical Activity Condition: Physically inactive older adults in this condition will perform 3 months of prescribed brisk walking (to increase cardio respiratory fitness) in their real world environments, using mobile health (mHealth) devices during each exercise session to achieve and maintain a minimum of 150 minutes of moderate to vigorous physical activity (MVPA) per week.
- Healthy Aging Education Condition: The education control condition will provide participants with materials and homework assignments on issues related to successful aging, such as nutrition, healthcare, and the typical changes associated with aging.
Period: Overall Study
Arm/Group | Physical Activity Condition | Healthy Aging Education Condition
Started | 21 | 23
Completed | 17 | 21
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Coronavirus (COVID)-19 shutdown | 0 | 1

BASELINE CHARACTERISTICS:
Population: In total, 44 participants were randomized to the intervention, with 21 in the Physical Activity Condition and 23 in the Healthy Aging Education Condition. One participant who was randomized to the Healthy Aging Education Condition could not finalize the baseline measurement appointment due to the COVID-19 pandemic shutting down research operations. Therefore, the analytical sample consisted of 43 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Activity Condition | Healthy Aging Education Condition | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.24 (4.27) | 72.27 (4.14) | 71.77 (4.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 16 | 21 | 37
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 22 | 40
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 22 | 43
Baseline MVPA [Mean (Standard Deviation); unit: Average MVPA minutes per day] — Average daily minutes spent in moderate to vigorous physical activity (MVPA) was defined as accelerometer counts per minute >= 1952. Participants wore the accelerometer on the hip for one week while asked to continue performing their regular activities in their natural environment.
  Average MVPA minutes per day | 26.37 (17.31) | 21.32 (17.42) | 23.8 (17.36)

OUTCOME MEASURES:

1. Primary Outcome: Moderate to Vigorous Physical Activity (MVPA) Average Per Day
Description: Average minutes per day spent in moderate to vigorous levels of physical activity (MVPA) (defined as =>1952 accelerometer counts per minute). MVPA minutes were determined based on one-week of accelerometer wear on the hip at baseline and post intervention.
Time Frame: Pre (baseline) and post (3 months)
Population: All participants who were randomized and completed the baseline sessions were included in the analyses (N=43).
Measure: Mean (Standard Deviation); unit: average minutes per day
Arm/Group | Physical Activity Condition | Healthy Aging Education Condition
Number analyzed (Participants) | 21 | 22
average minutes per day
  Pre MVPA average minutes per day | 26.37 (17.31) | 21.34 (17.44)
  Post MVPA average minutes per day | 44.09 (25.28) | 25.28 (15.99)

2. Secondary Outcome: Cerebral Blood Flow (Hippocampal and Frontal)
Description: Average cerebral blood flow measured with arterial spin labeling magnetic resonance imaging in ml/100g/min. Cerebral blood flow was obtained via arterial spin labeling MRI and Freesurfer software was utilized to delineate regions of interest for each participant (right and left regions were averaged). For the frontal lobe cerebral blood flow we averaged the mean of superior frontal, rostral and caudal middle frontal, pars opercularis, pars triangularis, pars orbitalis, lateral and medial orbitofrontal, precentral, paracentral, and frontal pole.
Time Frame: Pre (baseline) and post (3 months)
Population: We provide descriptive statistics for pre and post cerebral blood flow in the hippocampus and frontal cortex.
Measure: Mean (Standard Deviation); unit: ml/100g/minute
Arm/Group | Mobile Health Walking Condition | Healthy Aging Education Condition
Number analyzed (Participants) | 21 | 22
ml/100g/minute
  Pre hippocampal cerebral blood flow | 40.4 (10.82) | 41.03 (12.24)
  Post hippocampal cerebral blood flow | 35.36 (5.56) | 40.99 (9.1)
  Pre frontal cerebral blood flow | 45.52 (11.58) | 47.24 (10.46)
  Post frontal cerebral blood flow | 41.31 (7.41) | 46.96 (10.7)

3. Other Pre Specified Outcome: Memory Function
Description: A memory composite score was created by converting raw scores into z-scores and then averaging them for the following tests: Rey Auditory Verbal Learning Test trials 1 to 5, trial 6 (short-delay free recall), and delayed recall; Wechsler Memory Scale - Revised Logical Memory I and II (immediate and delayed recall scores). Z-scores were calculated using raw scores for these tests in the entire sample [(raw score-mean of the sample)/standard deviation of the sample]. Z-scores of 0 represent the sample's mean performance on the tests, z-scores >0 indicate better performance compared to the sample's mean, while z-scores <0 indicate worse performance compared to the sample's mean.
Time Frame: Pre (baseline) and post (3 months)
Population: All participants completed neuropsychological testing at pre and post.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Physical Activity Condition | Healthy Aging Education Condition
Number analyzed (Participants) | 21 | 22
z-score
  Pre memory score | .08 (.8) | -.07 (.82)
  Post memory score | -.10 (.94) | .09 (.68)

4. Other Pre Specified Outcome: Executive Function
Description: An executive function composite score was created by converting raw scores into z-scores and then averaging them for the following tests: Trail Making Test Part B minus Trail Making Test Part A, Golden version of the Stroop Color Word Trial, and verbal fluency (letters F,A,S). Trail making test scores were reversed prior to averaging, so higher scores = better performance. Z-scores were calculated using raw scores for these tests in the entire sample [(raw score-mean of the sample)/standard deviation of the sample]. Z-scores of 0 represent the sample's mean performance on the tests, z-scores >0 indicate better performance compared to the sample's mean, while z-scores <0 indicate worse performance compared to the sample's mean.
Time Frame: Pre (baseline) and post (3 months)
Population: All participants were included and descriptive statistics are presented for pre and post.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Physical Activity Condition | Healthy Aging Education Condition
Number analyzed (Participants) | 21 | 22
z-score
  Pre executive function score | .15 (.69) | -.14 (.80)
  Post executive function score | .07 (.73) | -.06 (.84)

5. Other Pre Specified Outcome: Cardiorespiratory Fitness
Description: Total time it takes the participant to reach 85% of their estimated maximal heart rate (220-age) measured via sub-maximal treadmill test in seconds.
Time Frame: Pre (baseline) and post (3 months)
Population: Descriptive data are presented for pre and post.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Physical Activity Condition | Healthy Aging Education Condition
Number analyzed (Participants) | 21 | 22
seconds
  Pre cardiorespiratory fitness (seconds) | 873.48 (175.47) | 840.55 (277.62)
  Post cardiorespiratory fitness (seconds) | 995.71 (157.43) | 948.61 (172.52)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse events recording followed the National Institute on Aging (NIA) Adverse Event and Serious Adverse Event Guidelines as outlined by the study's Data and Safety Monitoring Plan (DSMP), which included a safety officer. All adverse events were carefully monitored via telephone contact throughout the trial and were reported to the Institutional Review Board (IRB) of the University of California, San Diego, and the NIA program official following National Institutes of Health (NIH) guidelines.
Arm/Group | Physical Activity Condition | Healthy Aging Education Condition
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 3/21 | 2/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Activity Condition (N=21) | Healthy Aging Education Condition (N=22)
Non serious adverse event (Renal and urinary disorders) | 1 (1) | 0 (0) — Participant had to undergo emergency surgery for a renal/urinary issue. Unrelated to the study
Non serious adverse event (Eye disorders) | 1 (1) | 0 (0) — Participant reported experiencing blurry vision while at home. Not study related.
Non serious adverse event (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Back pain during treadmill walking at home.
Non serious adverse event (Social circumstances) | 0 (0) | 1 (1) — Participant tripped and scraped leg.
Non serious adverse event (Social circumstances) | 0 (0) | 1 (1) — Tripped during treadmill test.

LIMITATIONS AND CAVEATS:
Due to the COVID-19 pandemic, recruitment was terminated early, leading to a smaller than expected sample. As such, results are presented as descriptive statistics for pre and post intervention time points.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT03058146/Prot_SAP_000.pdf